## Preschooler Emotion Regulation in the Context of Maternal Borderline Personality Disorder Study Protocol NCT03060902

April 11, 2023

Initial phone screening was conducted to ensure that all mothers were biological mothers with at least 50% physical custody of the target child since birth. During this call, all mothers also completed the 10-item McLean Screening Instrument for Borderline Personality Disorder (MSI-BPD; Zanarini et al., 2003): scores ≥7 were required for the BPD groups and scores <2 were required for the HC group. In addition, mothers in the BPD group were asked about current treatment engagement and any mothers currently participating in DBT services were deemed ineligible. Eligibility was further determined during an in-person clinical intake, which included semi-structured diagnostic interviews for mothers. Trained research personnel administered the Structured Clinical Interview for the fifth edition of Diagnostic and Statistical Manual of Mental Disorders (DSM-5) (SCID-5; First, Williams, Karg, & Spitzer, 2016) and the Structured Interview for DSM-IV Personality (SIDP-IV; Pfohl, Blum, & Zimmerman, 1995) to determine eligibility. Approximately, 20% of intake interviews were double-coded from digital recordings and showed strong inter-rater reliability (Krippendorff's  $\alpha = .91$ ). Mothers in the BPD group met at least three diagnostic criteria for BPD, with one of these three symptoms being affective instability or uncontrolled anger. HC mothers reported no history of psychiatric illness (e.g., depression, anxiety) currently or since their child's conception, and showed no evidence of clinically significant ER difficulties as determined by scoring 0 on the affective instability and uncontrolled anger criteria on the SID-P. In addition, any mothers in a current psychotic or manic episode were deemed ineligible. All mothers and children also completed the Peabody Picture Vocabulary Test Fourth Edition (PPVT-IV; Dunn & Dunn, 2007) and the Expressive Vocabulary Test Second Edition (EVT-2; Williams, 1997) to provide an estimate of IQ. All eligible participants demonstrated standard scores ≥70. Eligible mothers who were in the BPD group were then randomized to receive DBT Skills or Family Services As Usual.

Those who were eligible were enrolled to complete four laboratory assessments (baseline, 4-month, 8-month, and 12-month followups). This assessment schedule paralleled the 12-month DBT treatment schedule (described below). Assessments were conducted by research assistants blinded to mother's group status and included questionnaires to assess maternal ER and behavioral tasks that assessed each of the four child ER domains (described below). Mothers also provided contact information for their child's preschool teacher or daycare provider. Following the baseline and 12-month laboratory assessment, teachers or daycare providers were contacted and asked to complete an online questionnaire assessing internalizing and externalizing problems observed in the preschool/daycare setting.